CLINICAL TRIAL: NCT04121845
Title: The Influence of Coronary Sinus Reducer Implantation on Exertional Capacity, Extent of Myocardial Ischemia and hrECG Markers of Arrhythmogenicity in Patients With Refractory Angina Pectoris
Brief Title: CoROnary SinuS Reducer implantatiOn for ischemiA reDuction
Acronym: CrossRoad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matjaž Bunc, Head of catheterization laboratory, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CrossRoad
Record Dates: First submitted 2019-10-06; First posted 2019-10-10 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Refractory Angina Pectoris
Keywords: angina pectoris; coronary sinus reducer; quality of life; reversible ischemia; exercise testing; oxygen consumption
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Punction of the right internal jugular vein and CSR implantation procedure simulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Active Comparator): Coronary sinus reducer implantation through right internal jugular vein.
  Interventions: Device: Coronary Sinus Reducer device
- Sham group (Sham Comparator): Puncture of the right internal jugular vein and simulation of the CSR implantation procedure.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: Coronary Sinus Reducer device — Coronary sinus reducer device (Neovasc, Richomnd, Canada) implantation in the coronary sinus. The procedure is performed in the cardiac catheterization laboratory through right internal jugular vein.
  Arms: Treatment group
Other: Sham procedure — Puncture of the right internal jugular vein and simulation of the CSR implantation procedure.
  Arms: Sham group

SUMMARY:
Patients with refractory angina pectoris have low quality of life and reduced exertional capacity. Studies have shown that the coronary sinus reducer (CSR) implantation improves the quality of life. However, to date there are no firm objective data on improvement of exertional capacity. Studies have shown a large influence of placebo effect after interventional procedures, which is even more pronounced than in medically treated patients. As angina pectoris presents entirely subjective perception of chest discomfort, its improvement may be influenced by this effect in up to 30 %. The investigators will study weather the CSR implantation improves aerobic exertional capacity in comparison to optimal medical therapy alone. Further, the investigators will explore the extent of myocardial reversible ischemia reduction and possible influence on hrECG markers of left ventricular arrhythmogenicity. 40 patients with refractory angina CCS class (Canadian cardiovascular society) II-IV and confirmed reversible ischemia will be included. Patients will be randomized into two groups. The first group will undergo CSR implantation procedure. The second group will present a sham control group with placebo procedure. At inclusion and after 6 months the investigators will perform cardiopulmonary exercise test (CPET), single photon emission tomography for detection of reversible ischemia (SPECT), high resolution ECG (hrECG), echocardiography and asses the subjective burden of angina according to CCS score and the quality of life according to the Seattle angina Questionnaire (SAQ).

ELIGIBILITY:
Inclusion Criteria:

* angina pectoris CCS class II-IV
* receiving optimal medical therapy for at least one month
* confirmed reversible myocardial ischemia in left anterior descending coronary artery (LAD) and/or left circumflex coronary artery (LCX) territory by SPECT
* not candidate for percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)

Exclusion Criteria:

* recent non stable angina pectoris (within 1 months)
* recent acute coronary syndrome (within 3 months)
* recent successful PCI and/or CABG (within 6 months)
* decompensated heart failure and/or recent (within 3 months) hospitalization due to heart failure
* severe heart valve(s) disease
* advanced chronic obstructive pulmonary disease (COPD) or poorly managed asthma
* peripheral arterial disease, musculoskeletal disorder or central nervous system disease which preclude exercise testing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Impact of CSR versus placebo procedure on exertional capacity measured by maximal oxygen consumption (VO2) during cardio-pulmonary exercise testing. | 6 months
  Maximal oxygen consumption on cycle spiroergometry using the same ramp exercise protocol during the same part of the day.

SECONDARY OUTCOMES:
Impact of CSR versus placebo procedure on exercise duration time during cardio-pulmonary exercise testing. | 6 months
  Exercise duration time on cycle spiroergometry using the same continuous exercise protocol during the same part of the day.
Change in the extent of myocardial reversible ischemia calculated by single-photon emission computed tomography (dynamic scintigraphy). | 6 months
  Dynamic myocardial scintigraphy with the use of a 4 segment model of the left ventricle for calculation of absolute regional perfusion (ml/g/min) during rest and during pharmacologic stress. Change in the extent of myocardial reversible ischemia calculated by single-photon emission computed tomography.
Change in the extent of myocardial reversible ischemia calculated by single-photon emission computed tomography (static scintigraphy). | 6 months
  Static myocardial scintigraphy with the use of a 17 segment model for the relative calculation of regional perfusion during rest and pharmacologic stress.
Change in RR interval variability as assessed by hrECG. | 6 months
  5 min recording of hrECG (1000 Hz) for the calculation of RR interval variability.
Change in late potentials as assessed by hrECG. | 6 months
  5 min recording of hrECG (1000 Hz) for the calculation of late potentials.
Change in QT variability as assessed by hrECG. | 6 months
  5 min recording of hrECG (1000 Hz) for determination of QT variability.
Change in Canadian Cardiovascular Society angina pectoris class (CCS). | 3 months, 6 months
  Change in CCS class I-IV. Acco
Impact of CSR versus placebo procedure on quality of life according to Seattle angina questionnaire (SAQ). | 3 months, 6 months
  Change in each of the five categories: Physical Limitation Scale (range 1-100), Anginal Stability Scale (range 1-100), Anginal Frequency Scale (range 1-100), Treatment Satisfaction Scale (range 1-100), Disease Perception Scale (range 1-100). Higher values in scale represent better outcome. Subscales are not combined.

OTHER OUTCOMES:
Influence of CSR implantation on echocardiographically assessed left ventricular elastance. | 6 months
Influence of CSR implantation on diastolic strain. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matjaž Bunc, Prof., Principal Investigator — University Medical Centre Ljubljana, Slovenia; David Žižek, Assoc. Prof., Study Chair — University Medical Centre Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication All IPD on special request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study completion and results publication. Not limited.
Access Criteria: All IPD that underlie results in a publication on editor/researcher request. All IPD on special request.

REFERENCES:
- [Background] Mannheimer C, Camici P, Chester MR, Collins A, DeJongste M, Eliasson T, Follath F, Hellemans I, Herlitz J, Luscher T, Pasic M, Thelle D. The problem of chronic refractory angina; report from the ESC Joint Study Group on the Treatment of Refractory Angina. Eur Heart J. 2002 Mar;23(5):355-70. doi: 10.1053/euhj.2001.2706. No abstract available. PMID 11846493
- [Background] Henry TD, Satran D, Hodges JS, Johnson RK, Poulose AK, Campbell AR, Garberich RF, Bart BA, Olson RE, Boisjolie CR, Harvey KL, Arndt TL, Traverse JH. Long-term survival in patients with refractory angina. Eur Heart J. 2013 Sep;34(34):2683-8. doi: 10.1093/eurheartj/eht165. Epub 2013 May 12. PMID 23671156
- [Background] Giannini F, Aurelio A, Jabbour RJ, Ferri L, Colombo A, Latib A. The coronary sinus reducer: clinical evidence and technical aspects. Expert Rev Cardiovasc Ther. 2017 Jan;15(1):47-58. doi: 10.1080/14779072.2017.1270755. PMID 27935738
- [Background] Konigstein M, Verheye S, Jolicoeur EM, Banai S. Narrowing of the Coronary Sinus: A Device-Based Therapy for Persistent Angina Pectoris. Cardiol Rev. 2016 Sep-Oct;24(5):238-43. doi: 10.1097/CRD.0000000000000101. PMID 26886464
- [Background] Verheye S, Jolicoeur EM, Behan MW, Pettersson T, Sainsbury P, Hill J, Vrolix M, Agostoni P, Engstrom T, Labinaz M, de Silva R, Schwartz M, Meyten N, Uren NG, Doucet S, Tanguay JF, Lindsay S, Henry TD, White CJ, Edelman ER, Banai S. Efficacy of a device to narrow the coronary sinus in refractory angina. N Engl J Med. 2015 Feb 5;372(6):519-27. doi: 10.1056/NEJMoa1402556. PMID 25651246
- [Background] Konigstein M, Meyten N, Verheye S, Schwartz M, Banai S. Transcatheter treatment for refractory angina with the Coronary Sinus Reducer. EuroIntervention. 2014 Feb;9(10):1158-64. doi: 10.4244/EIJV9I10A196. PMID 24561732
- [Background] Abawi M, Nijhoff F, Stella PR, Voskuil M, Benedetto D, Doevendans PA, Agostoni P. Safety and efficacy of a device to narrow the coronary sinus for the treatment of refractory angina: A single-centre real-world experience. Neth Heart J. 2016 Sep;24(9):544-51. doi: 10.1007/s12471-016-0862-2. PMID 27299456
- [Background] Banai S, Ben Muvhar S, Parikh KH, Medina A, Sievert H, Seth A, Tsehori J, Paz Y, Sheinfeld A, Keren G. Coronary sinus reducer stent for the treatment of chronic refractory angina pectoris: a prospective, open-label, multicenter, safety feasibility first-in-man study. J Am Coll Cardiol. 2007 May 1;49(17):1783-9. doi: 10.1016/j.jacc.2007.01.061. PMID 17466229
- [Background] Myers J, Froelicher VF. Optimizing the exercise test for pharmacological investigations. Circulation. 1990 Nov;82(5):1839-46. doi: 10.1161/01.cir.82.5.1839. PMID 2225380
- [Background] Kralios AC, Nappi JM, Tsagaris TJ, Kralios FA, Kuida H. Paradoxical increase of ventricular fibrillation threshold in response to coronary sinus obstruction. Am Heart J. 1988 Feb;115(2):334-40. doi: 10.1016/0002-8703(88)90479-6. PMID 3341168
- [Background] Kralios AC, Anderson FL, Kralios FA. Protective effect of coronary sinus obstruction from primary ischemia-induced ventricular fibrillation in the dog. Am Heart J. 1993 Apr;125(4):987-95. doi: 10.1016/0002-8703(93)90105-i. PMID 8465771
- [Background] De Maria GL, Kassimis G, Raina T, Banning AP. Reconsidering the back door approach by targeting the coronary sinus in ischaemic heart disease. Heart. 2016 Aug 15;102(16):1263-9. doi: 10.1136/heartjnl-2016-309642. Epub 2016 Jun 10. PMID 27288281
- [Background] Baldetti L, Colombo A, Banai S, Latib A, Esposito A, Palmisano A, Giannini F. Coronary sinus Reducer non-responders: insights and perspectives. EuroIntervention. 2018 Feb 20;13(14):1667-1669. doi: 10.4244/EIJ-D-17-00626. PMID 29086709
- [Derived] Mrak M, Zlahtic T, Starc V, Ivanovski M, Bunc M, Zizek D. The Impact of Coronary Sinus Reducer on Arrhythmic Properties in Patients with Refractory Angina. Rev Cardiovasc Med. 2023 Dec 26;24(12):368. doi: 10.31083/j.rcm2412368. eCollection 2023 Dec. PMID 39077099